CLINICAL TRIAL: NCT02695017
Title: Comparison of Changes in Oxygen Saturation in Flywheel Exercise Versus Conventional Strength Machine
Brief Title: Changes in Oxygen Saturation in Two Exercise Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Daniel Muñoz-Garcia, Physiotherapist, Centro Universitario La Salle
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CSEULS-PI-086
Record Dates: First submitted 2016-02-08; First posted 2016-03-01 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Muscle Oxigenation; Strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iso inertial (Experimental): Subjects should do 12 exercise repetition with Iso inertial machine
  Interventions: Device: Iso inertial
- Conventional machine (Experimental): Subjects should do 12 exercise repetition with conventional machine
  Interventions: Device: Conventional machine

INTERVENTIONS:
Device: Iso inertial
  Arms: Iso inertial
Device: Conventional machine
  Arms: Conventional machine

SUMMARY:
The investigator will proceed to assess changes in oxygenation of muscle tissue, electromyographic activation and strength in healthy subjects. For this, a measurement of all demographic variables on the first day of the study as well as a familiarity with the equipment will be performed. Participants will start the intervention 48 hours later to proceed with the first intervention with one of the exercises in this research (inertial pulley or regular machine). Later on, 48 hours later participants will perform the latest intervention that has not yet done, thus generating a crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* No pain
* Non disease

Exclusion Criteria:

* Exercise experience

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Oxygen saturation of Vastus lateralis muscle during the exercise of each participant | one second
  physiological parameter (Percentage of local oxygen consume will be record in every stage of the investigation)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Muñoz, MSc, Principal Investigator — Centro La Salle Universitario
Locations (1):
- Centro Superior de Estudios Universitarios La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Research publication